CLINICAL TRIAL: NCT01875068
Title: Implementing a Program of Physician Supervision to Improve the Quality of Patient Referrals From Nurse Practitioners and Physician Assistants
Brief Title: A Program of Physician Supervision to Improve the Quality of Patient Referrals From Nurse Practitioners and Physician Assistants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit adequate numbers for study
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William C. Mundell, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-002913
Record Dates: First submitted 2013-06-03; First posted 2013-06-11 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Complex Patients
Keywords: referrals; nurse practitioners; physician assistants; consultative general internal medicine
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPs & PAs referral discussions with a supervising physician (Experimental): required consultations between NPs and PAs and their supervising physicians
  Interventions: Behavioral: Consultations between NPs and PAs and their supervising physicians
- NPs and PAs - no consultations with supervising physisians (Other): NPs and PAs who are not required to discuss patient referrals
  Interventions: Behavioral: versus NPs and PAs who are not required to discuss patient referrals (control group).

INTERVENTIONS:
Behavioral: Consultations between NPs and PAs and their supervising physicians — Required discussion with physician prior to referral by a nurse practitioner or physician assistant
  Arms: NPs & PAs referral discussions with a supervising physician
Behavioral: versus NPs and PAs who are not required to discuss patient referrals (control group).
  Arms: NPs and PAs - no consultations with supervising physisians

SUMMARY:
The investigators have previously demonstrated utilizing a validated tool, that the quality of referrals from nurse practitioners (NP) and physician assistants (PA) is less than referrals from physicians. The investigators hypothesize that with local physician input, the quality of referrals from nurse practitioners and physician assistants will improve. This is a prospective study comparing patient referrals from nurse practitioners and physician assistants with and without prior discussion with a local physician.

ELIGIBILITY:
All nurse practitioners and physician assistants in the Mayo Clinic Health System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Improved referrals from nurse practitioners and physician assistants to physicians as determined using a previously validated tool | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lohr, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials